CLINICAL TRIAL: NCT02809924
Title: Simulation-based Just-in-time Training for Teaching Neonatal Endotracheal Intubation: A Randomized Controlled Trial
Brief Title: Just-in-time Training for Teaching Neonatal Endotracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: Montreal Children's Hospital of the MUHC (Other); CHU de Quebec-Universite Laval (Other); Université de Sherbrooke (Other); Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Moussa, Neonatologist, Clinical assistant professor, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5443
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Intubation; Education; Simulation Training
Keywords: endotracheal intubation; teaching; just-in-time

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulation-based just-in-time training (Experimental): Viewing a short video showing the neonatal glottis of similar gestational age to the patient that is being intubated followed by practice on a mannequin (Laerdal® Neonatal Intubation Trainer, Laerdal Medical, Toronto, Canada) with supervision and feedback from a senior provider (low fidelity simulation).
  Interventions: Other: Simulation-based just-in-time training
- Video training (Active Comparator): 5 minutes video regarding endotracheal intubation
  Interventions: Other: Video training

INTERVENTIONS:
Other: Simulation-based just-in-time training — Video and low fidelity simulation (Laerdal® Neonatal Intubation Trainer, Laerdal Medical, Toronto, Canada)
  Arms: Simulation-based just-in-time training
Other: Video training — Video describing endotracheal intubation
  Arms: Video training

SUMMARY:
This study compares the use of simulation-based just-in-time training to video training in learning neonatal endotracheal intubation. Half of the participants will be trained using simulation-based just-in-time training and the other half using video training.

The hypothesis are

Primary hypothesis:

In the Neonatal Intensive Care Unit, use of simulation-based just-in-time training, compared to video training, will increase the rate of successful clinical endotracheal intubation by 20%.

Secondary hypotheses:

The investigators expect that simulation-based just-in-time training prior to clinical endotracheal intubation will decrease time to successful intubation and rate of endotracheal intubation related adverse events, namely mucosal trauma, oesophageal and endobronchial intubations. In addition, the investigators expect that simulation-based just-in-time training will increase residents' confidence level while performing clinical endotracheal intubation.

DETAILED DESCRIPTION:
The study will be a prospective randomized controlled trial, taking place in the NICU of CHU Sainte-Justine in Montréal, Quebec, Canada ; Montreal Children's Hospital of the MUHC, in Montreal, Quebec, Canada; CHU de Quebec-Universite Laval, CHU de Sherbrooke and the General Jewish Hospital.

Simulation-based just-in-time training

Simulation-based just-in-time training, completed before performing endotracheal intubation, will consist of viewing a short video showing the neonatal glottis of similar gestational age to the patient that is being intubated followed by practice on a mannequin (Laerdal® Neonatal Intubation Trainer, Laerdal Medical, Toronto, Canada) with supervision and feedback from a senior provider (low fidelity simulation). The videos of the neonatal glottises have been locally created, after parent consent, using live recordings of endotracheal intubations performed with the C-MAC videolarygnoscope (Karl Storz GmbH & Co. KG, Tuttlingen, Germany). The low fidelity simulation will be performed in situ in the physician meeting room in the neonatal intensive care unit. Senior providers will be instructed to also educate the resident to different aspects related to the procedure: indications, contraindications, anatomy, equipment, personnel, potential complications, appropriate aftercare and common pitfalls.

Video training

Residents will watch a 5 minutes video regarding endotracheal intubation, which covers the following topics: indications, contraindications, anatomy, equipment, personnel, procedural steps, potential complications, appropriate aftercare and common pitfalls.

Definitions

1. Intubation is a success if the endotracheal tube is placed in the trachea under the vocal cords. It is defined according to usual clinical norms: change in color of the carbon dioxide detector, vapour in the endotracheal tube, thoracic expansion, assessment of bilateral lung air entry, absence of air entry in the stomach by auscultation, and improvement of patient's clinical parameters: heart rate and arterial oxygen saturation.
2. Time to intubation is defined as the time from insertion of the laryngoscope blade in the patients' mouth until it is pulled out.
3. Oesophageal intubation is diagnosed when there is absence of clinical signs of a successful endotracheal intubation and possibly air entry in the stomach by auscultation.
4. Right bronchial main stem intubation is diagnosed on chest x-ray.
5. A trial is counted as an attempt if there has been insertion of the laryngoscope blade in the patient's mouth.

ELIGIBILITY:
Inclusion Criteria:

* All residents registered in the three first years of the general paediatrics program at University of Montreal, McGill University, University of Sherbrooke and University Laval will be approached to participate in the study.
* All endotracheal intubation procedures attempted by paediatric residents in the neonatal intensive care unit at CHU Sainte-Justine; at Montreal Children's Hospital of the MUHC; at CHU de Quebec-Universite Laval , at CHU de Sherbrooke and at General Jewish Hospital (McGill university) will be included in the study, regardless of the patient weight or gestational age.

Exclusion Criteria:

* Trainees: No exclusion criteria.
* Patients with major oral, cervical or upper airway malformations, urgent endotracheal intubations with the inability to prepare the Just-in-time training material, and an unexpected difficult endotracheal intubation (needing the assistance of the anaesthetist).

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Endotracheal intubation success rate | 5 minutes

SECONDARY OUTCOMES:
Time to successful intubation | 5 minutes
  Defined as the time from insertion of the laryngoscope blade in the patients' mouth until it is pulled out.
Endotracheal intubation related complications | 15 minutes
  mucosal trauma, oesophageal intubation and endobronchial intubation
Resident's level of confidence | 15 minutes
  survey

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Moussa, MD, Principal Investigator — St. Justine's Hospital
Locations (5):
- Canada (5):
  - Centre Hospitalier de l'Université Laval, Laval, Quebec
  - The Montreal Children's Hospital MUHC, Montreal, Quebec
  - CHU Sainte-Justine, Montreal, Quebec
  - General Jewish Hospital, Montreal, Quebec
  - Université de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gizicki E, Assaad MA, Masse E, Belanger S, Olivier F, Moussa A. Just-In-Time Neonatal Endotracheal Intubation Simulation Training: A Randomized Controlled Trial. J Pediatr. 2023 Oct;261:113576. doi: 10.1016/j.jpeds.2023.113576. Epub 2023 Jun 21. PMID 37353151